CLINICAL TRIAL: NCT04260542
Title: The Role of De Novo Lipogenesis in Regulation of Insulin Sensitivity in Adipose Tissue in Obese
Brief Title: De Novo Lipogenesis and Insulin Sensitivity in Obese
Acronym: DELISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Michaela Siklova, Deputy head of adipose tissue physiology lab, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NV19-01-00263
Record Dates: First submitted 2020-01-23; First posted 2020-02-07 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Insulin Resistance; Obesity
Keywords: adipose tissue; insulin resistance; obesity; ketogenic diet; de novo lipogenesis
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FAST Lean (Active Comparator): Short-term fasting (FAST), comparator group of lean subjects
  Interventions: Behavioral: Fasting/refeeding
- FAST Obese (Experimental): Short-term fasting (FAST), experimental group of obese subjects
  Interventions: Behavioral: Fasting/refeeding
- KETO Obese (Experimental): Medium-term ketogenic diet intervention (KETO), experimental group of obese subjects
  Interventions: Behavioral: Ketogenic diet/ fasting

INTERVENTIONS:
Behavioral: Fasting/refeeding — 2-days fasting followed by 2-days of refeeding. During the fasting period the subjects will be hospitalized to control their state of health and ensure fasting compliance. During refeeding the standardized meals will be provided to cover individual daily requirements (60% carbohydrates, 15% protein, 25 % fat).
  Other Names: FAST lean
  Arms: FAST Lean
Behavioral: Fasting/refeeding — 2-days fasting followed by 2-days of refeeding. During the fasting period the subjects will be hospitalized to control their state of health and ensure fasting compliance. During refeeding the standardized meals will be provided to cover individual daily requirements (60% carbohydrates, 15% protein, 25 % fat).
  Other Names: FAST obese
  Arms: FAST Obese
Behavioral: Ketogenic diet/ fasting — 1 month of fasting-mimicking ketogenic diet and subsequent 2-days of refeeding. The subjects will be instructed by nutritional specialist to follow isocaloric ketogenic diet consisting of 6% carbohydrates, 17 % of proteins and 77% fat to cover individual energy demand. During refeeding the standardized meals will be provided to cover individual daily requirements (60% carbohydrates, 15% protein, 25 % fat).
  Other Names: KETO obese
  Arms: KETO Obese

SUMMARY:
Disturbances of de novo lipogenesis (DNL) are one of the features of dysfunction of adipose tissue (AT). Disturbances of DNL play a role in development of metabolic complications of obesity. The goal of this project is to investigate novel pathways of DNL regulation. DNL will be studied during nutritional interventions in healthy and obese subjects in exposure to 2-days high carbohydrate diet preceded by a) 2-days fasting b) several weeks´ ketogenic diet. This nutritional protocol creates conditions for the study of prominent changes in DNL: suppression of DNL during fasting or ketogenic diet followed by stimulation during high-carbohydrate diet. Systemic phenotypic features and molecular indices of DNL regulation in AT will be followed during the protocols. Specific attention will be paid to newly reported pathway- hormone sensitive lipase and transcription factor ChREBP. The results will contribute to development of pharmacological approaches in the treatment of metabolic complications of obesity, targeted selectively to AT, without side effects in other tissues.

DETAILED DESCRIPTION:
The main goal of the proposed project is to characterize the regulation of de novo lipogenesis in AT, a pathway strongly associated with insulin sensitivity in humans. The project should provide information that will bring proof-of-concept for the development of AT DNL-targeting therapeutic strategies to decrease the metabolic risk in obese individuals. Two protocols in lean and obese women to modulate (inhibit/induce) DNL will be implemented: 1) two days of fasting followed by two days of high-carbohydrate diet refeeding (FAST/RF) in lean and obese women; 2) "fasting-mimicking" intervention in obese women with high fat low carbohydrate ketogenic diet followed by two days of high-carbohydrate diet refeeding (KETO/RF). KETO diet should provide long lasting AT DNL inhibition, and as such it should further highlight the processes necessary for DNL activation in the refeeding phase. The unique protocols proposed in the application will allow to investigate in humans the relationship between AT DNL and whole body insulin sensitivity and glucose tolerance. Moreover, the state of the art experimental methodologies applied for the analyses of AT samples should uncover the possible mechanisms of regulation of DNL by ChREBP, HSL and other factors as well as the related AT secretory capacity in humans. The findings obtained in lean subjects will be compared to obese subjects, as the deregulated response of these pathways might be expected. The project will provide a proof-of-principle for the role of AT DNL in the regulation of insulin sensitivity in lean and obese individuals. The results will indicate novel pathways for future development of drugs targeting the relevant sites in AT in the context of treatment of obesity-induced insulin resistance and associated disorders.

ELIGIBILITY:
Inclusion Criteria:

* sedentary premenopausal women
* lean (n=20-25, age 25-40 years, BMI 20-25 kg/m2)
* obese (n=20-25, age 25-40 years, BMI 30-40 kg/m)

Exclusion Criteria:

* diagnosed cancer
* diabetes (T1DM and T2DM)
* liver and renal diseases
* major cardiovascular event
* bariatric surgery
* allergy to lidocaine
* positive serology for hepatitis (B and C) and HIV
* smoking above 10 cigarettes/day, alcohol consumption above 66g/day
* sleep apnea
* poor venous status
* weight-change more than 3kg in last 3 months
* untreated hyper- or hypo-thyroidism
* long term use of medication and/or steroids
* shift workers and individuals with abnormal sleep/wake pattern

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | through study completion, an average of 1 year
  Change in insulin sensitivity index (ΔiAUC insulin/ΔiAUC glucose from OGTT)
De Novo Lipogenesis in adipose tissue | through study completion, an average of 1 year
  Change in mRNA expression of lipogenic genes and by targeted and non-targeted lipid analysis (ΔCT)

SECONDARY OUTCOMES:
gene expression profiling of adipose tissue | through study completion, an average of 1 year
  Change in long non-coding RNA analysis by microarrays (ΔCT)

OTHER OUTCOMES:
Exploratory outcome into adipose tissue lipolysis | through study completion, an average of 1 year
  Change in glycerol, FFA concentration in AT explants
Exploratory outcome into liver lipogenesis | through study completion, an average of 1 year
  Change in amount of liver fat and VLDL-TG composition

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Siklova, PhD, Principal Investigator — Charles University, Czech Republic
Locations (2):
- Czechia (2):
  - Charles University, Prague
  - Faculty Hospital Kralovske Vinohrady, Prague